CLINICAL TRIAL: NCT07038005
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of SPGL008 Monotherapy for Patients With Advanced Malignant Tumors
Brief Title: A Phase I Study of SPGL008 in Subjects With Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Collaborators: Shenzhen Sciprogen Bio-pharmaceutical Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPGL008-101
Record Dates: First submitted 2025-06-17; First posted 2025-06-26 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Advanced Malignant Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- dose level 1 of SPGL008 （Intravenous administration） (Experimental)
  Interventions: Drug: SPGL008
- dose level 2 of SPGL008 （Intravenous administration） (Experimental)
  Interventions: Drug: SPGL008
- dose level 3 of SPGL008 （Intravenous administration） (Experimental)
  Interventions: Drug: SPGL008
- dose level 4 of SPGL008 （Intravenous administration） (Experimental)
  Interventions: Drug: SPGL008
- dose level 5 of SPGL008 （Intravenous administration） (Experimental)
  Interventions: Drug: SPGL008
- dose level 6 of SPGL008 （Intravenous administration） (Experimental)
  Interventions: Drug: SPGL008
- dose level 7 of SPGL008 （Intravenous administration） (Experimental)
  Interventions: Drug: SPGL008
- dose level 8 of SPGL008 （Intravenous administration） (Experimental)
  Interventions: Drug: SPGL008
- dose level 1 of SPGL008 （Subcutaneous administration） (Experimental)
  Interventions: Drug: SPGL008
- dose level 2 of SPGL008 （Subcutaneous administration） (Experimental)
  Interventions: Drug: SPGL008
- dose level 3 of SPGL008 （Subcutaneous administration） (Experimental)
  Interventions: Drug: SPGL008
- dose level 4 of SPGL008 （Subcutaneous administration） (Experimental)
  Interventions: Drug: SPGL008
- dose level 5 of SPGL008 （Subcutaneous administration） (Experimental)
  Interventions: Drug: SPGL008
- dose level 6 of SPGL008 （Subcutaneous administration） (Experimental)
  Interventions: Drug: SPGL008

INTERVENTIONS:
Drug: SPGL008 — Biological product

SUMMARY:
This study includes two cohorts, respectively evaluating safety, tolerability and preliminary efficacy of intravenous and subcutaneous administration of SPGL008.

DETAILED DESCRIPTION:
This study is a study of SPGL-008 monotherapy in patients with advanced malignant tumors. The study includes two cohorts, Cohort 1 and Cohort 2 will be administered by intravenous and subcutaneous administration respectively. Both cohorts will be conducted by the dose-escalation design to evaluate safety, tolerability and preliminary efficacy of different administration of SPGL008.

ELIGIBILITY:
Inclusion Criteria:

1. Males and/or females, 18-75 years old;
2. Histologically and/or cytologically documented advanced or metastatic malignant Tumors;
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
4. Expected survival >=3 months;
5. Signed informed consent form.

Exclusion Criteria:

1. Known uncontrolled or symptomatic central nervous system metastatic disease;
2. Adverse events (with exception of alopecia and fatigue) from any prior anticancer therapy of grade >1 (National Cancer Institute Common terminology Criteria [NCI-CTCAE] v.5.0);
3. Inadequate organ or bone marrow function;
4. Pregnant or breast-feeding woman;
5. Known allergies, hypersensitivity, or intolerance to SPGL008.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-09-22 (Estimated); Study Completion 2027-06-08 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | During the first cycle. Each cycle is 21 days
  DLT will be defined as toxicities that meet pre-defined severity criteria(according to the NCI CTCAE v5.0 toxicity assessment criteria), and assessed as having a suspected relationship to study drug that occurred within the first cycle(21 days) of treatment.
Maximum tolerated dose (MTD) | During the first cycle. Each cycle is 21 days
  MTD was defined as the highest dose at which dose-limiting toxicity (DLT) occurred in less than 33% of patients.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years
  Defined as the percentage of Complete Response (CR) plus partial response (PR) assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria.
Cmax | Up to 2 years
Tmax | Up to 2 years
T1/2 | Up to 2 years
AUC | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No